CLINICAL TRIAL: NCT00834054
Title: Interest of Repeated Extravascular Lung Water Measurements With the PICCO Device in Lung Transplanted Patients
Brief Title: Measurement of Lung Water by Transpulmonary Thermodilution in Lung Transplanted Patients
Acronym: PICCO-LungT
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2008/18
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Mucoviscidosis; Pulmonary Insufficiency
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Double-lung transplanted patients
  Interventions: Procedure: Double-lung transplantation

INTERVENTIONS:
Procedure: Double-lung transplantation — Double-lung transplanted patients

SUMMARY:
Repeated measurements of lung water by single transpulmonary thermodilution during the first postoperative days following lung transplantation

ELIGIBILITY:
Inclusion Criteria:

* double-lung transplanted patients

Exclusion Criteria:

* none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: double-lung transplanted patients
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
extra-vascular lung water | first postoperative days

SECONDARY OUTCOMES:
pulmonary permeability index | first postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Charles Cerf, MD, Study Chair — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France